Effect of transversus abdominis plane block combined with general anesthesia on perioperative stress response in patients undergoing radical gastrectomy

NCT number: NCT03035916

2017.1.30

## Statistical Analysis Plan

Based on a pilot study, we estimated the minimum detectable difference of plasma concentration of cortisol immediately after surgery among three groups. Through analysis by PASS 11.0 (NCSS Statistical Software, Kaysville, UT), at lease 25 participants each arm were needed. Taking into account the withdrawal of patients in the middle of the study, each group were more than a few included.

Data were stored in a Microsoft Office Excel 2007 spreadsheet and all statistical analyses were performed with SPSS (*ver.18.0, Chicago, IL, USA*). Parametric values were expressed as mean (SD), median (range), or percentages of the total number of patients (%). Thereafter, we used 1-way analysis of variance (ANOVA) and 2-tailed Dunnett test for pain scores, NE, E, Cor, cytokines, and hemodynamic data when compared among different groups. Categorical data were analyzed by using χ2 or Fisher exact test as appropriate. Levene test was used for homogeneity of variances. P value <0.05 was considered significant.